CLINICAL TRIAL: NCT03815812
Title: A Randomized, Double-blind, Placebo-controlled, Repeated-dosing, Multiple Ascending Dose Trial to Evaluate the Safety and Tolerability of a Novel PCSK-9 Anti-body, IBI306, in Chinese Patients With Hypercholesterolemia
Brief Title: Multiple Ascending Dose Study of PCSK-9 Inhibitor (IBI306) in Chinese Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI306B101
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI306 (Experimental): Participants received one of 6 dose levels of IBI306 administered as multiple subcutaneous dose
  Interventions: Drug: IBI306
- placebo (Placebo Comparator): Participants received matching placebo dose regimen by subcutaneous injection.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IBI306 — Cohort 1: 75mg Q2W Cohort 2: 140mg Q2W Cohort 3: 300mg Q4W Cohort 4: 420mg Q4W Cohort 5: 450mg Q6W Cohort 6: 600mg Q6W
  Arms: IBI306
Drug: placebo — Cohort 1: 75mg Q2W Cohort 2: 140mg Q2W Cohort 3: 300mg Q4W Cohort 4: 420mg Q4W Cohort 5: 450mg Q6W Cohort 6: 600mg Q6W
  Arms: placebo

SUMMARY:
IBI306 is a fully human monoclonal antibody that binds proprotein convertase substilisin/kexin type 9 (PCSK-9), preventing its interaction with the low-density lipoprotein cholesterol receptor (LDL-R) and thereby restoring LDL-R recycling and low-density lipoprotein cholesterol（LDL-C）uptake. In phase I study IBI306 was shown to be safe and well tolerated. There was robust reduction in LDL-C, Apo(B), non-HDL-C and lipoprotein (a) in healthy subjects. This study is a randomized, double-blind, placebo-controlled, repeated-dosing, multiple ascending dose trial to evaluate the safety and tolerability of a novel PCSK-9 anti-body, IBI306, in Chinese patients with hypercholesterolemia.

DETAILED DESCRIPTION:
A total of 60 patients who meet the criteria for admission and have a clinical diagnosis of hypercholesterolemia and have received statin for at least 4 weeks will be randomized and receive different dose groups of IBI306 or matching placebo. Ascending dose design includes 6 dose levels: 75 mg Q2W, 140 mgQ2W, 300 mg Q4W，420mg Q4W, 450 mg Q6W，and 600 mg Q6W. Total duration of the study per subject is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria in order to be included in the study:

  * Provide a signed and dated informed consent form;
  * Men or women with an age of 18 to 70 years of age at screening (Inclusive);
  * BMI between18kg/m2 and 30kg/m2(Inclusive);
  * Diagnosis of hyperlipidemia, and taking statins with moderate doses or above for at least 4 weeks;
  * Fasting LDL-C between 100 mg / dl (2.6 mmol / L) and 220 mg / dl (5.7 mmol / L) at screening (Inclusive);
  * Fasting triglycerides ≤ 400 mg (4.5 mmol / L) at screening.

Exclusion Criteria:

* Subjects who do not meet any of the following exclusion criteria cannot be included in the study:

  * Subject's current statin treatment are stable less than 4 weeks prior to random enrollment
  * New York Heart Association (NYHA) III or IV heart failure, or last left ventricular ejection fraction <30%
  * Uncontrolled hypertension, defined as repeated measurements confirmed, sitting systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg.
  * Diabetic patients have one of the following conditions;

    1. Known microvascular and macrovascular complications
    2. HbA1c>7.5% within 4 weeks before screening
  * Moderate or severe renal insufficiency, defined as the estimated glomerular filtration rate <60 ml / min / 1.73 m2 during screening (calculated using the MDRD formula)
  * Active liver disease or impaired liver function, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the normal upper limit (ULN) at screening.
  * Have previously undergone liver transplant surgery.
  * Creatine kinase (CK) ≥ 3 times the upper limit of normal (ULN) at screening.
  * At the discretion of the investigator, there are known active infections or major blood, kidney, metabolism, gastrointestinal or endocrine dysfunction.
  * Female subject of childbearing potential not willing to use an acceptable method(s) of effective birth control during treatment with investigational product and for an additional 15 weeks after the end of treatment with investigational product. Male subjects are reluctant to inform their female sexual partners about their participation in the clinical study.
  * Female subject is pregnant or breast feeding, planning to become pregnant or planning to breastfeed during treatment with investigational product and/or within 15 weeks after the end of treatment with investigational product..
  * Subjects have been treated with PCSK9 inhibitors or have participated in other PCSK-9 inhibitor studies
  * Subject has known sensitivity to the study drug and its excipients
  * Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment (for example, alcohol or other substance abuse, unable or unwilling to comply with the agreement or mental illness).
  * Currently receiving treatment in another investigational device or drug study, or less than 30 days before randomization since ending treatment on another investigational device or drug study(s) while participating in this study
  * In the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
AEs/SAEs | up to 12 weeks
  • Percentage of participants with adverse events and severity of adverse events from the first dose to the last visit

SECONDARY OUTCOMES:
Tmax | up to 12 weeks
Cmax | up to 12 weeks
area under curve (AUC) | up to 12 weeks
volume of distribution (Vd) | up to 12 weeks
half-life (T1/2) | up to 12 weeks
clearance (CL) | up to 12 weeks
accumulation factor (AR) | up to 12 weeks
changes in blood PCSK-9 concentrations at different time points before and after administration relative to baseline | up to 12 weeks
ADA | up to 12 weeks
  The occurrence of anti-IBI306 antibody (ADA) in serum before and after administration
NAb | up to 12 weeks
  The occurrence of neutralizing antibody (NAb) in serum before and after administration
Percent change in LDL-C from baseline at 12 weeks | baseline and week 12
Changes in LDL-C levels from baseline at 12 weeks | baseline and week 12
Percent change in non-HDL-C cholesterol levels from baseline at 12 weeks | baseline and week 12
Percent change in ApoB from baseline at 12 weeks | baseline and week 12
Percent change in ApoB/ApoA1 ratio from baseline at 12 weeks | baseline and week 12
Percent of patients with a 15% or more decrease in LDL-C levels from baseline at 12 weeks | baseline and week 12
Percent change in Lp(a) from baseline at 12 weeks | baseline and week 12
Percent change in mean LDL-C levels at week 6 and 12 relative to baseline | baseline, week 6 and 12
Percent change in mean ApoB levels at week 6 and 12 relative to baseline | baseline, week 6 and 12
Percent change in mean Lp(a) levels at week 6 and 12 relative to baseline | baseline, week 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Cui, Principal Investigator — Peking University First Hospital; Huo Yong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui Y, Zhao X, Qi L, Li X, Huang Z, Yang G, Qian L, Deng H, Li H, Huo Y. A Potential Long-Acting LDL-Cholesterol-Lowering PCSK9 Monoclonal Antibody: Randomized, Placebo-Controlled Phase 1 Studies. JACC Asia. 2021 Nov 9;1(3):411-415. doi: 10.1016/j.jacasi.2021.09.002. eCollection 2021 Dec. PMID 36341216